CLINICAL TRIAL: NCT07334769
Title: Religiously Integrated Cognitive Behavioral Group Therapy for Generalized Anxiety Disorder
Brief Title: Religiously Integrated Cognitive Behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Haldun University (Other)
Responsible Party: Principal Investigator, Dilek Ekinci, Clinical Psychologist, Ibn Haldun University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-71395021-020-9865
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-01

CONDITIONS: Anxiety Disorder (Panic Disorder or GAD); Well Being
Keywords: generalized anxiety disorder; group therapy; cognitive behavioral group therapy; well-being
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Generalized Anxiety Disorder

STUDY DESIGN:
Masking Description: This study is open-label. Due to the nature of the psychological group interventions, neither participants nor therapists could be blinded to treatment allocation. Outcome measures were based on self-report scales.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional Cognitive Behavioral Group Therapy (Active Comparator): Participants in this group received 10 sessions of online cognitive behavioral group therapy
  Interventions: Behavioral: Traditional Cognitive Behavioral Group Therapy
- Waiting Group (Other): There is no intervention for this group
  Interventions: Other: Waiting Group
- Religiously Integrated Cognitive Behavioral Group Therapy (Experimental): Participants in this group received 10 sessions of online religiously integrated cognitive behavioral group therapy
  Interventions: Behavioral: Religiosly Integrated Cognitive Behavioral GroupTherapy

INTERVENTIONS:
Behavioral: Religiosly Integrated Cognitive Behavioral GroupTherapy — This intervention consists of a structured, group-based, online cognitive behavioral therapy program integrated with participants' spiritual/religious values. The program includes psychoeducation about anxiety, cognitive restructuring, exposure to uncertainty, problem-solving, and behavioral exercises, combined with spiritually framed coping strategies such as meaning-making, patience, gratitude, trust, and values-based reflection. Sessions were delivered weekly in a standardized manualized format by a trained therapist. The intervention aimed to reduce anxiety symptoms and enhance psychological well-being.
  Arms: Religiously Integrated Cognitive Behavioral Group Therapy
Behavioral: Traditional Cognitive Behavioral Group Therapy — his intervention consists of a structured, group-based, online cognitive behavioral therapy program focusing on anxiety management. The program includes psychoeducation, cognitive restructuring, graduated exposure to anxiety-provoking situations and intolerance of uncertainty, problem-solving, and behavioral exercises. Sessions were delivered weekly in a standardized, manualized format by a trained therapist, without spiritual or religious content.
  Arms: Traditional Cognitive Behavioral Group Therapy
Other: Waiting Group — Participants assigned to the waitlist control group did not receive any active intervention during the study period and were offered the intervention after completion of post-test assessments.
  Arms: Waiting Group

SUMMARY:
This study aims to examine the effect of a newly developed religously oriented cognitive behavioral group therapy program on the level of anxiety and well-being in young adults compared to the traditional cognitive behavioral therapy-based program.

Hypoteses 1 Religiously oriented CBT group therapy will be more effective in reducing participants' general anxiety levels compared to traditional CBT group therapy and the control group, and this effect will continue in the two-month follow-up measurements.

Hypoteses 2 Religiously oriented CBT group therapy will be more effective in increasing participants' levels of well-being compared to traditional CBT group therapy and the control group, and this effect will continue in the two-month follow-up measurements.

ELIGIBILITY:
Inclusion Criteria:

Being between 18 and 45 years of age, Willingness to participate in 10 weekly group sessions, Having a GAD-7 score of 5 or higher, Exhibiting symptoms of generalized anxiety disorder as determined by the Structured Clinical Interview for DSM-5 (SCID-5-CV), Having regular access to the internet.

Exclusion Criteria:

Currently receiving any form of psychological treatment Having previously undergone long-term psychotherapy Having a primary comorbid psychological disorder other than generalized anxiety disorder, Expressing suicidal ideation, Having completed only primary school education

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Anxiety | Baseline (pre-test), immediately post-intervention (post-test), and 2-month follow-up.
  The Anxiety Thoughts Inventory (AnTI) is a self-report measure assessing the frequency of anxiety-related thoughts. The total score is calculated by summing item responses, with higher scores indicating greater levels of maladaptive anxious thinking. Lower scores reflect fewer anxiety-related cognitions and improvement over time. Change in scores from baseline to post-intervention and follow-up represents a reduction in anxiety-related thought patterns.

SECONDARY OUTCOMES:
Well-being | Baseline (pre-test), immediately post-intervention (post-test), and 2-month follow-up.
  The PERMA Well-Being Scale is a self-report measure assessing overall psychological well-being across five domains: Positive Emotion, Engagement, Relationships, Meaning, and Accomplishment. Total scores are derived by averaging item responses, with higher scores indicating higher levels of psychological well-being. An increase in total score reflects improvement in overall well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Ekinci, PhD Candidate, Principal Investigator — Ibn Haldun University
Locations (1):
- İstanbul, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data (IPD) will be made available beginning 6 months after publication of the primary study results and will remain available for a period of 5 years.

DOCUMENTS (1):
  • Study Protocol (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT07334769/Prot_000.pdf